CLINICAL TRIAL: NCT03263975
Title: Effects of Dehydration on Neuromuscular Performance and Sympathetic Control of Cardiovascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-03H
Record Dates: First submitted 2017-08-23; First posted 2017-08-28 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Dehydration Hypertonic; Isotonic Dehydration
MeSH Terms: interventions — gatorade

STUDY DESIGN:
Intervention Model Description: Between groups design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise heat STress (EHS) (Experimental): EHS - dehydration produced by sweating and fluid restriction; primary loss of body water accompanied by small loss of electrolytes (hypertonicity). Interventions include rehydration with Gatorade or Enterade oral rehydration therapies.
  Interventions: Other: Gatorade or Enterade
- Lasix (LAS) (Experimental): LAS - dehydration produced by Lasix (diuretic, 80 mg oral dose) administration to produce losses of body water accompanied by large losses of electrolytes (isotoncity). Interventions include rehydration with Gatorade or Enterade oral rehydration therapies.
  Interventions: Other: Gatorade or Enterade

INTERVENTIONS:
Other: Gatorade or Enterade — Commercially available oral rehydration therapies

SUMMARY:
The mechanism(s) by which dehydration (both intra- and extracellular) impairs performance are still poorly described. A loss of volume results in increased occurrence of orthostatic intolerance, including dizziness, fatigue, headaches and related symptoms with upright posture. Any of these symptoms can contribute to decreased performance in maneuvers performed in the upright posture, which includes many military tasks. Thus, loss of volume challenges the cardiovascular and blood pressure responses to systemic whole body endurance exercise, while osmolality is the stimulus for intracellular dehydration that may impair local muscle force production by impairing contractile function, neural signaling, or both. In this study, we will compare how both types of dehydration affect MSNA and CAC.

The results of this study will provide mechanistic insight for how dehydration (intra- or extracellular) impairs systemic whole body and local small muscle performance in vivo. This Basic Science study seeks to understand how volume and osmolality impact MSNA and CAC as a basis for improving potential countermeasures, such as a more optimally formulated rehydration beverage. Therefore, this study directly complements Task Area T10 (Hot Weather Operations and Hydration: Injury and Performance Optimization) and impacts virtually all 14 Military Operational Medicine Research Program Drivers.

DETAILED DESCRIPTION:
Study Objectives and Hypotheses

Primary Objective

The primary objectives of this study are to understand the in vivo effects of dehydration on:

1. Sympathetic neural control of cardiovascular function (MSNA), and
2. Neuromuscular function (CAC) via the IT Test

The primary hypotheses of this study are:

1. Baseline MSNA, and MSNA responses to tilt, will be higher in response to extracellular dehydration due to larger intravascular volume losses and greater baroreceptor unloading.
2. Neuromuscular function (CAC) via the IT Test will a) be more impaired by intracellular dehydration (cell stress) and b) CAC will show a greater performance reduction than CAR because it reduces the emphasis placed on the voluntary portion of performance (i.e., MVC).

Ancillary Questions/Sub Studies

1. The collection of blood and urine before and after exercise-heat stress and dehydration provides an opportunity to measure and characterize cytokine and intestinal barrier integrity marker (I-FAB, claudin-3) responses (blood) and renal stress biomarkers (urine) in humans. This descriptive research 'sub-study' directly complements Task Area T10 (Hot Weather Operations and Hydration: Injury and Performance Optimization) near and mid-term research goals of identifying biomarkers of heat stress for protection against heat injury. There are no hypotheses associated with this sub-study.
2. The study of dehydration requires rehydration for recovery. Rehydration provides an opportunity for a novel comparison of renal water retention (urine volume) when consuming equal volumes of two different commercial beverages (Gatorade® or Enterade-S®). Unlike Gatorade®, which is a carbohydrate-based beverage containing electrolytes, Enterade-S® is an amino acid-based beverage containing electrolytes. We hypothesize that the unique formulation of Enterade-S® will improve the rate of fluid absorption and fluid retention compared to Gatorade® in both intracellular and extracellular dehydration trials.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-45
* In good health as determined by OMSO General Medical Clearance
* Passed his/her most recent Army Physical Fitness Test (APFT) (military volunteers only) or exercise at least 2 times per week (civilian volunteers)
* Ability to comprehend and willingness to sign informed consent

Exclusion Criteria:

* Females who are pregnant or planning to become pregnant during the study
* Taking prescription or over the counter medication, other than a contraceptive (unless approved by OMSO and PI)
* Physical problems/injuries associated with walking or cycling
* Allergy to sulfa drugs (Lasix™ or sulfonamide antibiotics such as Septra™)
* Allergy to skin adhesive
* Hemoglobinopathy (sickle cell trait)
* Heart, lung, kidney, muscle, or nerve disorder(s)
* History of heat or orthostatic intolerance
* Diagnosed and/or treated for fluid/electrolyte imbalance within the last 30 days
* Presence of metal implants/electronic medical devices in lower extremities
* Current or previous (within the past 5 years) diagnosis of any autonomic disorder, including idiopathic orthostatic intolerance, orthostatic hypotension, postural tachycardia syndrome (POTS), or neurocardiogenic syncope (MSNA group only)
* Tobacco/nicotine use (MSNA group only)
* Significant muscle, joint, or bone injury affecting the legs within the last 6 months (CAC group only)
* Difficulty swallowing large pills
* History of obstructive disease of the gastrointestinal tract including (but not limited to) diverticulosis, diverticulitis and inflammatory bowel disease, peptic ulcer disease, Crohn's disease, ulcerative colitis; or previous gastrointestinal surgery.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2016-12-08 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Water and electrolyte retention | 180 minutes
  Mass balance measures of total body water and electrolytes

SECONDARY OUTCOMES:
Body water compartment changes | 180 minutes
  Osmometric measurements and calculations of body fluid spaces

IPD SHARING:
Plan to Share IPD: No